CLINICAL TRIAL: NCT03163576
Title: The Efficacy and Safety of Niacin on Hyperphosphatemia in End Stage Renal Disease Patients Undergoing Haemodialysis
Brief Title: The Efficacy of Niacin on Hyperphosphatemia in Patients Undergoing Haemodialysis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, EYAbdelhafez, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENPD
Record Dates: First submitted 2017-05-21; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — Niacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): patients received niacin 750 mg twice daily up to 2000 mg in addition to usual phosphate binders .
  Interventions: Drug: Niacin; Drug: Phosphate Binder
- control group (Active Comparator): patients received usual phosphate binders .
  Interventions: Drug: Phosphate Binder

INTERVENTIONS:
Drug: Niacin — tablets
  Arms: study group
Drug: Phosphate Binder — tablets

SUMMARY:
Hyperphosphatemia is a common complication of end-stage renal disease and particularly affects haemodialysis patients. Elevated serum phosphorus contributes to the development of secondary hyperparathyroidism, Mineral bone disorders,metastatic calcifications and calcific uremic arteriolopathy. There is a significant association between hyperphosphatemia and increased morbidity and mortality in end stage renal disease patients including cardiovascular morbidity and mortality ,also it's associated with hospitalization of haemodialysis patients.

DETAILED DESCRIPTION:
Hyperphosphataemia is mainly due to impaired renal phosphate excretion and primary increase in renal phosphate reabsorption,due to acute or chronic renal insufficiency. Renal excretion is so efficient in normal subjects that balance can be maintained with only a minimal rise in serum phosphorus concentration even for a large phosphorus load. Therefore, acute hyperphosphataemia usually resolves within few hours if renal function is intact.

Although, there is multiple lines of treatment of hyperphosphatemia in end stage renal disease patients undergoing Hemodialysis but still inadequate. As Calcium containing phosphate binders may sometimes result in adverse effects such as hypercalcemia. Non-calcium containing phosphate binders, such as sevelamer and lanthanum, are expensive. Aluminum-containing agents are efficient but no longer widely used because of their toxicity. Several trials have shown that nicotinamide and niacin are capable of remarkably reducing serum phosphate levels in patients undergoing haemodialysis.

Niacin is a water-soluble vitamin, and a part of the B complex vitamin, both nicotinamide and niacin (nicotinic acid) are forms of vitamin B3 . As a broad-spectrum drug that can affect lipid levels, niacin reduces levels of total cholesterol, triglyceride, and low-density lipoprotein cholesterol, while increasing high-density lipoprotein cholesterol levels. Niacin also lowers serum phosphorus levels in patients with chronic kidney disease, dyslipidemia, and diabetes mellitus. Furthermore, niacin plays a key role in cardiovascular diseases and cardiovascular-related mortality by modifying both dyslipidemia and phosphorus levels.

Recently, nicotinic acid and related compounds such as nicotinamide have also been shown to decrease phosphorus absorption in the gastro-intestinal tracts of animals by a different mechanism than the traditional phosphate binders.

The major side effects of niacin are vasodilation and flushing, which appear to be mediated through prostaglandin production, and thus can be attenuated by premedication with aspirin.

ELIGIBILITY:
Inclusion Criteria:

1. end stage renal disease patients aged from 18-60 years old.
2. Duration of Hemodialysis >6 months.
3. Serum phosphorus level >5 mg/dl

Exclusion Criteria:

* 1)patients on sevelamer or cinacalcet. 2)Hepatitis C virus +ve patients. 3)Connective tissue disease. 4)Active malignancy. 5) pregnancy 6) active peptic ulcer disease 7) treatment with carbamazepine.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
the level of phosphorous level in haemodialysis patients treated by niacin | two years
  laboratory test

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rennick A, Kalakeche R, Seel L, Shepler B. Nicotinic acid and nicotinamide: a review of their use for hyperphosphatemia in dialysis patients. Pharmacotherapy. 2013 Jun;33(6):683-90. doi: 10.1002/phar.1258. Epub 2013 Mar 21. PMID 23526664
- [Background] Lenglet A, Liabeuf S, Guffroy P, Fournier A, Brazier M, Massy ZA. Use of nicotinamide to treat hyperphosphatemia in dialysis patients. Drugs R D. 2013 Sep;13(3):165-73. doi: 10.1007/s40268-013-0024-6. PMID 24000048
- [Background] Edalat-Nejad M, Zameni F, Talaiei A. The effect of niacin on serum phosphorus levels in dialysis patients. Indian J Nephrol. 2012 May;22(3):174-8. doi: 10.4103/0971-4065.98751. PMID 23087550
- [Background] Jin Kang H, Kim DK, Mi Lee S, Han Kim K, Hee Han S, Hyun Kim K, Eun Kim S, Ki Son Y, An WS. Effects of low-dose niacin on dyslipidemia and serum phosphorus in patients with chronic kidney disease. Kidney Res Clin Pract. 2013 Mar;32(1):21-6. doi: 10.1016/j.krcp.2012.12.001. Epub 2012 Dec 31. PMID 26889433
- [Background] Malberti F. Hyperphosphataemia: treatment options. Drugs. 2013 May;73(7):673-88. doi: 10.1007/s40265-013-0054-y. PMID 23625273
- [Background] Zahed NS, Zamanifar N, Nikbakht H. Effect of low dose nicotinic acid on hyperphosphatemia in patients with end stage renal disease. Indian J Nephrol. 2016 Jul-Aug;26(4):239-43. doi: 10.4103/0971-4065.161020. PMID 27512294
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086